CLINICAL TRIAL: NCT02867228
Title: Noninvasive Estimation of Work of Breathing
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Resources to be able to screen and enroll patients are no longer available.
Sponsor: Respironics, California, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-AAAP8801
Record Dates: First submitted 2016-08-10; First posted 2016-08-15 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2016-08

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Observational Group (Other): Patients receiving mechanical ventilation and subject to the intervention: changes in ventilator settings.
  Interventions: Other: changes in ventilator settings

INTERVENTIONS:
Other: changes in ventilator settings — Ventilator settings will be adjusted (vent mode, pressure support/control level, cycling, inspiratory time, mandatory rate).

SUMMARY:
This study will evaluate the correlation between invasively measured parameters (work of breathing/power of breathing, resistance and elastance), derived using esophageal pressure measurements, and their corresponding non-invasive estimated values (noninvasive work of breathing/power of breathing, resistance and elastance), computed using airway pressure and flow measurements only.

DETAILED DESCRIPTION:
This study will evaluate the correlation between invasively measured parameters (work of breathing/power of breathing, resistance and elastance), derived using esophageal pressure measurements, and their corresponding non-invasive estimated values (noninvasive work of breathing/power of breathing, resistance and elastance), computed using airway pressure and flow measurements only. Vent settings will be adjusted to test accuracy over a range of respiratory support conditions.

ELIGIBILITY:
Inclusion Criteria:

* Adult medical/surgical ICU patients (Age≥18) on mechanical ventilation for respiratory failure, spontaneously breathing and receiving eligible for pressure support ventilation (PSV).

Exclusion Criteria:

* Prisoners and patients with closed-head injury (e.g., trauma), hemodynamic instability, multiple organ system failure or late term pregnancy will not be studied.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-05-04 (Actual); Study Completion 2017-05-04 (Actual)

PRIMARY OUTCOMES:
Accuracy of lung mechanics measurements | Immediate

CONTACTS AND LOCATIONS:
Overall Officials: David H Chong, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Banner MJ, Kirby RR, Kirton OC, DeHaven CB, Blanch PB. Breathing frequency and pattern are poor predictors of work of breathing in patients receiving pressure support ventilation. Chest. 1995 Nov;108(5):1338-44. doi: 10.1378/chest.108.5.1338. PMID 7587438
- [Result] Kirton OC, DeHaven CB, Hudson-Civetta J, Morgan JP, Windsor J, Civetta JM. Re-engineering ventilatory support to decrease days and improve resource utilization. Ann Surg. 1996 Sep;224(3):396-402; discussion 402-4. doi: 10.1097/00000658-199609000-00016. PMID 8813268